CLINICAL TRIAL: NCT02837432
Title: The Effect of Cortisol Administration on Neural Correlates of Emotion in Depression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Keith Sudheimer, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19771
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Depression
Keywords: Depression; Cortisol; Sadness; Genetics; Stress
MeSH Terms: conditions — Depression | interventions — hydrocortisone acetate; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy (Other): Healthy individuals will receive both the placebo and hydrocortisone interventions in a randomized order
  Interventions: Drug: Hydrocortisone acetate; Drug: Placebo
- Depression (Other): Individuals with depression will receive both the placebo and hydrocortisone interventions in a randomized order
  Interventions: Drug: Hydrocortisone acetate; Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone acetate
  Other Names: Cortef
Drug: Placebo

SUMMARY:
There is good evidence to suggest that the pathological version of sadness that people with Major Depression experience could be caused by the failure of the hormone cortisol to properly inhibit sadness-related brain activity in the subgenual cingulate cortex. This project investigates if the subgenual cingulate cortex has become insensitive to cortisol in patients with depression and tests for variants of the cortisol receptor genes that could predispose individuals to develop cortisol insensitivity.

ELIGIBILITY:
https://redcap.stanford.edu/surveys/?s=3F7WCENPND

Inclusion Criteria:

* Healthy Participants must have no Axis 1 mental disorder
* Participants with depression must meet minimum severity levels (Hamilton >7)
* All participants must weight less than 280 pounds for the purposes of MRI scanning

Exclusion Criteria:

In order to protect against risk associated with taking Hydrocortisone, all participants must not have any of the following:

* Psychotropic medications
* Recent surgery
* Endocrine disorders
* Liver disease
* Kidney disease
* Thyroid disorder
* History of malaria
* Tuberculosis
* Osteoporosis
* Glaucoma/cataracts
* Chronic expressed infections (herpes --including ocular herpes, HIV, etc.)
* History of congestive heart failure
* History of recurring seizures
* Stomach Ulcers
* Comorbid psychosis
* Current use of illicit drugs
* High Blood pressure

In order to protect against risks associated with MRI scanning participants must not be/have any of the following:

* >280 lbs
* In-dwelling ferrous metals
* Left Handed
* Abnormal Hearing
* Claustrophobic
* Head injury with loss of consciousness

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Sadness-induced subgenual cingulate activity as measured by functional magnetic resonance imaging. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sudheimer, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Department of Psychiatry and Behavioral Sciences, 401 Quarry Road, Stanford, California, United States